CLINICAL TRIAL: NCT01224067
Title: A Double-Blind, Placebo-Controlled, Flexible-Dosage Study to Evaluate the Efficacy and Safety of Adjunctive Quetiapine in the Treatment of Refractory Social Anxiety Disorder in Adults
Brief Title: Adjunctive Quetiapine in the Treatment of Refractory Social Anxiety Disorder in Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cambridge Health Alliance (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CHA-IRB-0094/11/04
Record Dates: First submitted 2010-09-10; First posted 2010-10-19 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Social Anxiety Disorder
MeSH Terms: conditions — Phobia, Social | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quetiapine (Active Comparator): Quetiapine (dosage 50mg to 300mg + sertraline)Experimental
  Interventions: Drug: Quetiapine
- Placebo (Placebo Comparator): Participant will receive placebo for 8 weeks.
  Interventions: Drug: Quetiapine

INTERVENTIONS:
Drug: Quetiapine — Adjunctive quetiapine -Participant will receive up to 300 mg/day of quetiapine for 8 weeks.
  Other Names: Seroquel

SUMMARY:
This is a 16-week research study in which participants suffering from Social Anxiety Disorder (SAD) will receive Sertraline (a medication FDA approved for the treatment of SAD) for the first 8 weeks. If a participant remains symptomatic, he/she will enter the second phase of the study in which he/she continues taking Sertraline but also randomly receives either Seroquel or placebo in conjunction with Sertraline for additional 8 weeks. The purpose of this study is to determine the efficacy of adjunctive Seroquel in treating SAD.

DETAILED DESCRIPTION:
This will be a single-site study aimed at evaluating the safety, tolerability, and efficacy of quetiapine as compared to placebo in the treatment of generalized anxiety disorder. This will be an 8-week open-label sertraline trial followed by a randomized double-blind placebo-controlled, parallel-group prospective study. Participants will first receive sertraline (25-200 mg/day) for 8 weeks. Patients who remain symptomatic - are considered refractory - and meet inclusion criteria will be randomized and enter the double-blind phase. They will receive either adjunctive quetiapine (25-400 mg/day) or placebo for 8 weeks. The primary outcome measures are change in the Liebowitz Social Anxiety Scale(LSAS) and Clinical Global Impression of Improvement (CGI-I) scores. The proposed sample size is 80 subjects. Patients will be discontinued from the study if needed due to ineffectiveness or excessive side effects. Measurements of changes in efficacy and side effects will be carried out every weekly visit. Enrollment will occur over 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients, age 18-65.
* Diagnosis of Social Anxiety Disorder (SAD), generalized subtype, by DSM-IV criteria.
* Liebowitz Social Anxiety Scale (LSAS) rating greater than or equal to 50 for both phases.
* Hamilton Depression Scale (HAM-D-17) score less than or equal to 16.

Exclusion Criteria:

* Pregnant or lactating women or others not using acceptable means of birth control (e.g., IUD, oral contraceptives, barrier devices, condoms and foam, implanted progesterone rods stabilized for at least 3 months).
* Patients with current or history of bipolar disorder, schizophrenia, or other psychotic conditions.
* Patients with a history of alcohol or substance abuse or dependence within the last six months or a positive toxicology screen consistent with abuse at baseline.
* Patients with significant unstable medical illness, including any medical pathology considered not well-controlled with conventional treatment, i.e., that may require during the study period medication adjustment, ongoing tests or procedures, intensive treatment or hospitalization. In addition, baseline laboratory tests will be conducted and required to be within normal limits or have no clinical significance for patient entry in the study.
* Severe personality disorders likely to interfere with study participation or who, in the investigator's judgment, pose a current, serious suicidal or homicidal risk.
* Ongoing psychotherapy directed toward the treatment of social anxiety disorder.
* History of hypersensitivity to sertraline and quetiapine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-03; Primary Completion 2008-07 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Liebowitz Social Anxiety Scale (LSAS) | Change from Baseline to Endpoint at 8 weeks
  Change from Baseline to Endpoint of social anxiety symptoms after 8 weeks of treatment. Assessed weekly throughout the study for a total of 8 weeks.

SECONDARY OUTCOMES:
Clinical Global Impression of Improvement (CGI-I) scores | Change from Baseline to Endpoint at 8 weeks
  Change from Baseline to Endpoint after 8 weeks of treatment in overall clinical improvement of social anxiety symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo D Kinrys, MD, Principal Investigator — Cambridge Health Alliance; Harvard Medical School
Locations (1):
- Cambridge Health Alliance, Cambridge, Massachusetts, United States